CLINICAL TRIAL: NCT02759146
Title: Using SMART Design to Improve Symptom Management Strategies Among Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Gwen Wyatt, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PA13-165; R01CA193706 (NIH)
Record Dates: First submitted 2016-04-21; First posted 2016-05-03 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Reflexology (Experimental): Reflexology is a specialized foot therapy that applies a firm walking motion pressure to the feet. It is based on the premise that the foot has reflexes that mirror the rest of the body. It has been shown to reduce symptoms.
  Interventions: Other: Reflexology
- Meditative Practice (Experimental): Meditative Practices include elements of meditation, gentle yoga and breathing exercises. These practices focus purposeful attention to the present moment and have been shown to enhance one's ability to adapt to serious health concerns
  Interventions: Other: Meditative Practices
- Control (No Intervention): Control - no intervention

INTERVENTIONS:
Other: Reflexology — Reflexology is a specialized foot therapy that applies a firm walking motion pressure to the feet. It is based on the premise that the foot has reflexes that mirror the rest of the body. It has been shown to reduce symptoms.
  Arms: Reflexology
Other: Meditative Practices — Meditative Practices include elements of meditation, gentle yoga and breathing exercises. These practices focus purposeful attention to the present moment and have been shown to enhance one's ability to adapt to serious health concerns
  Arms: Meditative Practice

SUMMARY:
The purpose of this study is to compare reflexology to meditative practices to reduce symptoms in cancer patients.

DETAILED DESCRIPTION:
First, dyads were randomized to receive caregiver-delivered reflexology or meditative practice. Fatigue severity was assesses weekly via phone calls to the cancer patients during weeks 1-4 of the intervention. For patients who did not respond to the intervention during the first 4 weeks, those dyads were referred to as non-responder and re-randomized. A non-responder was determined if the level of reported fatigue remained the same or increased from the first week of the intervention.

The re-randomization placed the non-responders in either a group that received a higher dose (more time) with the first intervention or to the alternate practice (meditative practice to those randomized to reflexology and vice versa) for weeks 5-8. Those who did respond during weeks 1-4 continued the same therapy they began with.

ELIGIBILITY:
Inclusion Criteria:

* 21 year of age or older
* Solid tumor cancer diagnosis
* Able to perform basic activities of daily living (ADLs)
* Undergoing chemotherapy, hormonal therapy, or targeted therapy
* Able to speak and understand English
* Have access to a telephone
* Able to hear normal conversation
* Reporting a severity of 3 or higher on fatigue using a 0-10 standardized scale at intake.

Exclusion Criteria:

* Diagnosis of major mental illness on the medical record (verified by the recruiter)
* Residing in a nursing home
* Bedridden
* Currently receiving reflexology or meditative practices
* Suspected or diagnosed deep vein thrombosis or painful foot neuropathy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Wyatt, PhD, RN, Principal Investigator — Michigan State University College of Nursing
Locations (7):
- United States (7):
  - Arizona Oncology, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - Northwestern University, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - MSU Breslin Cancer Center, Lansing, Michigan
  - Sparrow Cancer Center, Lansing, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Findings from this study will be available to other researchers under the following conditions: 1) appropriate human subjects protection is in place; 2) data have been de-identified; and 3) study investigators have publicly presented and published key findings.

REFERENCES:
- [Derived] Thana K, Sikorskii A, Lehto R, Guhaniyogi P, Brewer S, Victorson D, Pace T, Badger T, Wyatt G. Family caregivers of those with cancer: quality of life outcomes from a sequential multiple assignment randomized trial. Support Care Cancer. 2022 Jul;30(7):5891-5902. doi: 10.1007/s00520-022-07012-7. Epub 2022 Apr 5. PMID 35378595

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 8 clinical centers between April 2015 and November 2019.
Pre-assignment Details: Of the 471 consented, 347 completed the baseline interview and were randomized. Between the time of consent and baseline interview 124 dyads attrited. Reasons included:
  Changed mind about participating (n=24), cannot be reached via phone/mail (n=55), too busy (n=19), too overwhelmed (n=8), too sick (n=9) and other reasons (n=48).
  Throughout the study, if either patient or caregiver dropped from the study, the dyad was considered an attrition.
Groups:
- Reflexology With Response, Then Continued Reflexology: Reflexology is a specialized foot therapy that applies a firm walking motion pressure to the feet. It is based on the premise that the foot has reflexes that mirror the rest of the body. It has been shown to reduce symptoms.
  Participants were randomized into the reflexology intervention, then after week 4 of symptom responses, were considered responders. Participants then continued with the reflexology intervention.
- Reflexology Non-responders, Then Continued Reflexology: Reflexology is a specialized foot therapy that applies a firm walking motion pressure to the feet. It is based on the premise that the foot has reflexes that mirror the rest of the body. It has been shown to reduce symptoms.
  Participants were randomized into the reflexology intervention, then after 4 weeks of symptom responses were considered non-responders. Participants then continued with the reflexology intervention.
- Reflexology Non-responders, Then Switch to Meditation: Reflexology is a specialized foot therapy that applies a firm walking motion pressure to the feet. It is based on the premise that the foot has reflexes that mirror the rest of the body. It has been shown to reduce symptoms.
  Meditative Practices include elements of meditation, gentle yoga and breathing exercises. These practices focus purposeful attention to the present moment and have been shown to enhance one's ability to adapt to serious health concerns.
  Participants were randomized into the reflexology intervention, then after 4 weeks of symptom responses were considered non-responders. Participants then switched to a meditative practice intervention.
- Meditative Practice With Response, Continued Meditation: Meditative Practices include elements of meditation, gentle yoga and breathing exercises. These practices focus purposeful attention to the present moment and have been shown to enhance one's ability to adapt to serious health concerns.
  Participants were randomized into the meditative practice intervention, then after 4 weeks of symptom response were considered responders. Participants then continued with the meditative practice intervention.
- Meditative Practice Non-responders, Continued Meditation: Meditative Practices include elements of meditation, gentle yoga and breathing exercises. These practices focus purposeful attention to the present moment and have been shown to enhance one's ability to adapt to serious health concerns.
  Participants were randomized into the mindfulness meditation intervention, then after 4 weeks of symptom responses were considered non-responders. Participants then continued with the meditative practice intervention.
- Meditative Practice Non-responders, Switch to Reflexology: Meditative Practices include elements of meditation, gentle yoga and breathing exercises. These practices focus purposeful attention to the present moment and have been shown to enhance one's ability to adapt to serious health concerns.
  Reflexology is a specialized foot therapy that applies a firm walking motion pressure to the feet. It is based on the premise that the foot has reflexes that mirror the rest of the body. It has been shown to reduce symptoms.
  Participants were randomized into the meditative practice intervention, then after 4 weeks of symptom responses were considered non-responders. Participants then switched to a reflexology intervention.
Period: Week 1-4
Arm/Group | Reflexology With Response, Then Continued Reflexology | Reflexology Non-responders, Then Continued Reflexology | Reflexology Non-responders, Then Switch to Meditation | Control | Meditative Practice With Response, Continued Meditation | Meditative Practice Non-responders, Continued Meditation | Meditative Practice Non-responders, Switch to Reflexology
Started (150 reflexology dyads, 150 mediative practice dyads, and 47 control dyads were randomized. Between the randomization and response to weekly calls, 24 reflexology dyads, 44 meditative practice dyads and 3 control dyads attrited from the study totaling n=71 attrited dyad between the start of participant flow. In the analysis of repeated measures, participants with at least one non-missing post-baseline value were included.) | 57 | 36 | 33 | 44 (One control participant could continue without the other after baseline.) | 49 | 30 | 27
Completed | 56 | 34 | 32 | 44 | 49 | 29 | 26
Not Completed | 1 | 2 | 1 | 0 | 0 | 1 | 1
Period: Week 5-8
Arm/Group | Reflexology With Response, Then Continued Reflexology | Reflexology Non-responders, Then Continued Reflexology | Reflexology Non-responders, Then Switch to Meditation | Control | Meditative Practice With Response, Continued Meditation | Meditative Practice Non-responders, Continued Meditation | Meditative Practice Non-responders, Switch to Reflexology
Started (In the analysis of repeated measures, participants with at least one non-missing post-baseline value were included. For example, if a participant dropped out before week 5 but completed one of the weeks 1-4, their data were included in the analysis of weeks 1-4 under the missing at random assumption. Same applies to the analysis of longitudinal data for weeks 5-12.) | 56 | 34 | 32 | 44 | 49 | 29 | 26
Completed (In the reflexology and meditative practices groups created by the first randomization, one participant could not continue without the other at week 5 unless the patient was a responder and dyad was not re-randomized.) | 46 | 29 | 22 | 37 | 44 | 23 | 20
Not Completed | 10 | 5 | 10 | 7 | 5 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Reflexology Patients: Patients randomized into the reflexology arm, given reflexology from a friend/ family member.
  Reflexology is a specialized foot therapy that applies a firm walking motion pressure to the feet. It is based on the premise that the foot has reflexes that mirror the rest of the body. It has been shown to reduce symptoms.
- Meditative Practice Patients: Patients randomized into the meditative practice arm, given meditative practice from a friend/ family member.
  Meditative Practices include elements of meditation, gentle yoga and breathing exercises. These practices focus purposeful attention to the present moment and have been shown to enhance one's ability to adapt to serious health concerns
- Control Patients: Control- no intervention
- Reflexology Caregivers: Caregivers providing reflexology to their friend/ family member.
  Reflexology is a specialized foot therapy that applies a firm walking motion pressure to the feet. It is based on the premise that the foot has reflexes that mirror the rest of the body. It has been shown to reduce symptoms.
- Meditation Practice Caregivers: Caregivers providing meditative practice to their friend/ family member.
  Meditative Practices include elements of meditation, gentle yoga and breathing exercises. These practices focus purposeful attention to the present moment and have been shown to enhance one's ability to adapt to serious health concerns
- Control Caregivers: Control - no intervention
- Total: Total of all reporting groups
Arm/Group | Reflexology Patients | Meditative Practice Patients | Control Patients | Reflexology Caregivers | Meditation Practice Caregivers | Control Caregivers | Total
Number analyzed (Participants) | 150 | 150 | 47 | 150 | 150 | 47 | 694
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Baseline measure separated by patient/ caregiver
  years
    Age- Caregiver: number analyzed (Participants) | 0 | 0 | 0 | 146 | 146 | 47 | 339
    Age- Caregiver |  |  |  | 56.07 (14.84) | 55.56 (14.58) | 54.59 (13.42) | 55.65 (14.50)
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Baseline measure separated by patient/ caregiver
  years
    Age- Patient: number analyzed (Participants) | 150 | 150 | 47 | 0 | 0 | 0 | 347
    Age- Patient | 56.65 (13.91) | 58.41 (12.29) | 59.31 (13.99) |  |  |  | 57.77 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participant did not respond
  Participants
    number analyzed (Participants) | 150 | 150 | 47 | 140 | 137 | 45 | 669
    Female | 116 | 115 | 34 | 84 | 76 | 26 | 451
    Male | 34 | 35 | 13 | 56 | 61 | 19 | 218
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participant did not respond
  Participants
    Race: number analyzed (Participants) | 150 | 150 | 47 | 139 | 145 | 47 | 678
    Race: White Caucasian | 126 | 129 | 46 | 119 | 119 | 40 | 579
    Race: Asian | 7 | 2 | 1 | 4 | 5 | 4 | 23
    Race: Black or African American | 12 | 12 | 0 | 8 | 12 | 0 | 44
    Race: Other | 5 | 7 | 0 | 8 | 9 | 3 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participant did not respond
  Participants
    Ethnicity: number analyzed (Participants) | 147 | 148 | 46 | 145 | 147 | 47 | 680
    Ethnicity: Hispanic | 23 | 7 | 3 | 17 | 7 | 3 | 60
    Ethnicity: Non Hispanic | 122 | 140 | 43 | 126 | 139 | 44 | 614
    Ethnicity: Other | 2 | 1 | 0 | 2 | 1 | 0 | 6
Number of comorbid conditions [Mean (Standard Deviation); unit: Number of conditions] — Population: Not all participants responded to question
  Number of conditions
    Comorbid conditions- patient: number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    Comorbid conditions- patient | 3.89 (2.83) | 3.83 (2.73) | 4.19 (3.35) |  |  |  | 3.90 (2.86)
    Comorbid conditions- caregiver: number analyzed (Participants) | 0 | 0 | 0 | 146 | 148 | 47 | 341
    Comorbid conditions- caregiver |  |  |  | 3.45 (2.56) | 2.93 (2.71) | 3.06 (2.54) | 3.17 (2.63)
Patient-caregiver relationship [Count of Participants; unit: Participants] — Population: Participant did not respond
  Participants
    number analyzed (Participants) | 145 | 147 | 47 | 145 | 147 | 47 | 678
    Spouse | 85 | 94 | 30 | 85 | 94 | 30 | 418
    Adult Child | 14 | 11 | 3 | 15 | 16 | 7 | 66
    Parent | 15 | 16 | 7 | 14 | 11 | 3 | 66
    Friend | 19 | 17 | 5 | 19 | 17 | 5 | 82
    Other | 12 | 9 | 2 | 12 | 9 | 2 | 46
Living arrangement [Count of Participants; unit: Participants] — Population: Not all patients/ caregivers responded
  Participants
    number analyzed (Participants) | 142 | 147 | 47 | 142 | 147 | 47 | 672
    Together | 100 | 112 | 34 | 100 | 112 | 34 | 492
    Separately | 42 | 35 | 13 | 42 | 35 | 13 | 180
Number of Complimentary and Alternative Medicine (CAM) therapies used [Mean (Standard Deviation); unit: Number of CAM therapies] — Population: Participants did not respond
  Number of CAM therapies
    number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    (all) | 2.36 (2.41) | 2.51 (2.23) | 2.00 (1.91) |  |  |  | 2.38 (2.27)
Education [Count of Participants; unit: Participants]
  High school or less | 2 | 4 | 0 | 25 | 18 | 6 | 55
  At least some college | 61 | 62 | 22 | 85 | 81 | 28 | 339
  Graduate/ professional degree | 45 | 33 | 11 | 36 | 49 | 13 | 187
Employment [Count of Participants; unit: Participants] — Population: Participant did not respond
  Participants
    number analyzed (Participants) | 147 | 146 | 47 | 145 | 147 | 47 | 679
    Employed full time | 46 | 44 | 13 | 78 | 67 | 18 | 266
    Employed part time | 9 | 15 | 4 | 11 | 15 | 5 | 59
    Retired | 9 | 6 | 2 | 42 | 47 | 16 | 122
    Not employed | 83 | 81 | 28 | 14 | 18 | 8 | 232
Income [Count of Participants; unit: Participants] — Population: Participant did not respond
  Participants
    number analyzed (Participants) | 146 | 148 | 46 | 134 | 137 | 43 | 654
    <= $24,000 | 18 | 8 | 1 | 13 | 9 | 4 | 53
    $25,000-$49,000 | 21 | 25 | 5 | 25 | 23 | 7 | 106
    $50,000-$99,000 | 30 | 28 | 7 | 32 | 42 | 6 | 145
    >=$100,000 | 17 | 24 | 11 | 24 | 20 | 11 | 107
    Other | 60 | 63 | 22 | 40 | 43 | 15 | 243
Brief Fatigue Inventory Severity of Fatigue (BFI, worst fatigue) [Mean (Standard Deviation); unit: units on a scale] — The BFI instrument consists of nine items. The first three items ask respondents to rate the severity of fatigue "right now," at its "usual" level during the past 24 hours and at its "worst" level during the past 24 hours. Answer choices are on a scale of 0 -10, where 0 = no fatigue and 10 = as bad as you can imagine. Higher score= worse outcome. Population: Caregivers did not report outcome measure
  units on a scale
    number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    (all) | 4.08 (2.90) | 3.95 (2.71) | 3.81 (2.63) |  |  |  | 3.99 (2.78)
Fatigue interference (BFI) [Mean (Standard Deviation); unit: units on a scale] — The second part of the BFI index The remaining six items assess how much fatigue interfered with: general activity, mood, walking ability, normal work (including work outside the home and daily chores), relations with other people, and enjoyment of life. Responses are on a 0 to 10 scale where 0=does not interfere and 10=completely interferes. High score= worse outcome. Population: Caregivers did not report outcome measure
  units on a scale
    number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    (all) | 20.14 (15.09) | 21.85 (16.14) | 21.91 (14.08) |  |  |  | 21.12 (15.40)
Summed severity of other symptoms (MDASI) [Mean (Standard Deviation); unit: units on a scale] — The expanded M.D. Anderson Symptom Inventory (MDASI) includes 19 symptoms: fatigue, pain, nausea, disturbed sleep, distress, shortness of breath, difficulty remembering, decreased appetite, drowsiness, dry mouth, sadness, vomiting, numbness/tingling, diarrhea, constipation, sore mouth, rash, hair loss, and cough, and the interference of these symptoms with daily life on the scale from 0 = symptom not present to 10 = worst imaginable. Scores are summed, higher score= worse outcome. Population: Caregivers did not report outcome measure
  units on a scale
    number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    (all) | 38.61 (29.00) | 40.43 (28.24) | 37.23 (22.46) |  |  |  | 39.20 (27.81)
Symptom interference (MDASI) [Mean (Standard Deviation); unit: units on a scale] — The MDASI measures how much the symptoms have interfered with six daily activities:
  general activity, mood, work, relations with others, walking, and enjoyment of life.
  Interference is rated on a 0-10 numerical rating scale, 0 being "did not interfere" and 10 being "interfered completely." High=worse outcome Population: Caregivers did not report outcome measure
  units on a scale
    number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    (all) | 19.06 (15.46) | 19.69 (15.35) | 18.98 (14.91) |  |  |  | 19.32 (15.30)
Patient Reported Outcomes Measurement Information System (PROMIS) depression [Mean (Standard Deviation); unit: units on a scale] — Self report of depression for patient or caregiver. A score of 50 represents the mean or average of the reference population. A score of 60 means that the participant is one standard deviation above the reference population (standard deviation=10 units).
  Higher score = worse outcome. Population: Not all participants responded to question
  units on a scale
    PROMIS depression- Patient: number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    PROMIS depression- Patient | 53.67 (8.52) | 53.13 (8.39) | 55.26 (7.98) |  |  |  | 53.65 (8.39)
    PROMIS depression- Caregiver: number analyzed (Participants) | 0 | 0 | 0 | 146 | 148 | 47 | 341
    PROMIS depression- Caregiver |  |  |  | 47.14 (7.61) | 45.41 (6.45) | 46.87 (7.82) | 46.35 (7.19)
PROMIS anxiety [Mean (Standard Deviation); unit: units on a scale] — Self reported anxiety measure for patient or caregiver. A score of 50 represents the mean or average of the reference population. A score of 60 means that the participant is one standard deviation above the reference population (standard deviation=10 units).
  Higher score = worse outcome. Population: Not all participants responded
  units on a scale
    PROMIS anxiety- Patient: number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    PROMIS anxiety- Patient | 54.34 (9.17) | 53.64 (8.66) | 55.01 (7.78) |  |  |  | 54.13 (8.76)
    PROMIS anxiety- Caregiver: number analyzed (Participants) | 0 | 0 | 0 | 146 | 147 | 47 | 340
    PROMIS anxiety- Caregiver |  |  |  | 48.38 (8.31) | 46.09 (7.67) | 48.10 (9.43) | 47.35 (8.26)
Attentional function index [Mean (Standard Deviation); unit: units on a scale] — The Attentional Function Index (AFI) is a self-report questionnaire consisting of 13 items on which respondents rate their effectiveness of their function on common tasks requiring attention and cognitive control from 0 (not at all) to 10 (extremely well).
  Scores are the average of all 13 items, high score= better outcome. Population: Caregivers did not report outcome information
  units on a scale
    Subscale 1 (action): number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    Subscale 1 (action) | 6.08 (2.22) | 6.19 (2.11) | 5.71 (2.45) |  |  |  | 6.08 (2.20)
    Subscale 2 (lapses): number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    Subscale 2 (lapses) | 3.50 (2.20) | 3.19 (2.25) | 3.21 (2.07) |  |  |  | 3.33 (2.20)
    Subscale 3 (effectiveness): number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    Subscale 3 (effectiveness) | 5.93 (1.71) | 6.04 (1.67) | 5.70 (1.93) |  |  |  | 5.95 (1.73)
Long Term Quality of Life (LTQL) spirituality [Mean (Standard Deviation); unit: units on a scale] — Spiritual/philosophical views of life subscale. Response range 0-44, higher is better. Population: Caregivers did not report outcome measure
  units on a scale
    number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    (all) | 34.27 (8.56) | 33.63 (7.30) | 33.26 (8.33) |  |  |  | 33.85 (7.99)
Social Support (MSPSS) [Mean (Standard Deviation); unit: units on a scale] — Measures perceived social support from different sources (family member or friend) based on a 12 item questionnaire, with a seven point response. 1=very strongly disagree, 7=very strongly agree. Response range 4-28, higher is better. Population: Caregivers did not report outcome measure
  units on a scale
    number analyzed (Participants) | 148 | 148 | 47 | 0 | 0 | 0 | 343
    (all) | 25.93 (4.46) | 26.40 (4.19) | 25.64 (3.07) |  |  |  | 26.09 (4.18)
PROMIS physical function [Mean (Standard Deviation); unit: units on a scale] — Self report of general physical functioning. A score of 50 represents the mean or average of the reference population. A score of 60 means that the participant is one standard deviation above the reference population (standard deviation=10 units).
  Higher score = better functioning. Population: Not all participants responded to question
  units on a scale
    PROMIS physical function- Patient: number analyzed (Participants) | 146 | 145 | 47 | 0 | 0 | 0 | 338
    PROMIS physical function- Patient | 39.97 (7.99) | 40.17 (8.58) | 39.91 (7.01) |  |  |  | 40.05 (8.10)
    PROMIS physical function- Caregiver: number analyzed (Participants) | 0 | 0 | 0 | 145 | 148 | 46 | 339
    PROMIS physical function- Caregiver |  |  |  | 54.00 (6.03) | 53.33 (6.74) | 52.40 (8.54) | 53.49 (6.73)
PROMIS sleep disturbance [Mean (Standard Deviation); unit: units on a scale] — Self report of quality of sleep in the past 7 days. A score of 50 represents the mean or average of the reference population. A score of 60 means that the participant is one standard deviation above the reference population (standard deviation=10 units).
  Higher score = worse outcome. Population: Patients did not report outcome measure
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 146 | 147 | 47 | 340
    (all) |  |  |  | 47.09 (7.18) | 46.29 (8.27) | 47.86 (7.80) | 46.85 (7.75)
PROMIS fatigue [Mean (Standard Deviation); unit: units on a scale] — Self report of fatigue in the last seven days. PROMIS fatigue only applies to caregivers as part of PROMIS-29 Profile T-score range 33.-75.8, higher is worse. Population: Patients did not report outcome measure
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 146 | 147 | 47 | 340
    (all) |  |  |  | 47.10 (9.03) | 45.40 (8.57) | 48.43 (9.78) | 46.55 (8.99)
PROMIS pain interference [Mean (Standard Deviation); unit: units on a scale] — Measure the self-reported consequences of pain on relevant aspects of a person's life. A score of 50 represents the mean or average of the reference population. A score of 60 means that the participant is one standard deviation above the reference population (standard deviation=10 units).
  Higher score = worse outcome. Population: Patients did not report outcome measure
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 145 | 147 | 47 | 339
    (all) |  |  |  | 47.59 (7.67) | 47.18 (7.85) | 49.28 (8.75) | 47.65 (7.91)
PROMIS pain intensity [Mean (Standard Deviation); unit: units on a scale] — Self report of pain at its worse in the past seven days. Response range 0-10, 0= no pain, 10= worst imaginable pain. Higher score= worse outcome. Population: Patients did not report outcome measure
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 145 | 147 | 47 | 339
    (all) |  |  |  | 1.51 (1.86) | 1.29 (1.84) | 1.64 (1.94) | 1.43 (1.86)
Satisfaction with participation in social roles [Mean (Standard Deviation); unit: units on a scale] — PROMIS measure of adult satisfaction with participation in social roles, responses on a five point scale with 1=not at all- 5=very much. High score= better outcome. For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population. Population: Patients did not report outcome measure
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 146 | 148 | 47 | 341
    (all) |  |  |  | 54.63 (8.69) | 55.94 (7.92) | 53.15 (9.23) | 55.00 (8.47)
Caregiver burden [Mean (Standard Deviation); unit: units on a scale] — Measure including five subscales: impact of caregiving on schedule, caregiver's esteem, family support, impact on health, and impact on finances. Each question had a five point response scale, 1=strongly disagree- 5=strongly agree. High score= higher burden, worse outcome. Population: Participant did not respond
  units on a scale
    Subscale 1 (impact): number analyzed (Participants) | 0 | 0 | 0 | 146 | 148 | 47 | 341
    Subscale 1 (impact) |  |  |  | 2.46 (0.88) | 2.35 (0.90) | 2.63 (0.76) | 2.44 (0.88)
    Subscale 2 (esteem): number analyzed (Participants) | 0 | 0 | 0 | 146 | 148 | 47 | 341
    Subscale 2 (esteem) |  |  |  | 4.54 (0.44) | 4.54 (0.37) | 4.40 (0.46) | 4.52 (0.42)
    Subscale 3 (support): number analyzed (Participants) | 0 | 0 | 0 | 146 | 148 | 47 | 341
    Subscale 3 (support) |  |  |  | 1.70 (0.68) | 1.67 (0.75) | 1.84 (0.66) | 1.71 (0.71)
    Subscale 4 (health): number analyzed (Participants) | 0 | 0 | 0 | 146 | 148 | 47 | 341
    Subscale 4 (health) |  |  |  | 1.47 (0.68) | 1.40 (0.63) | 1.63 (0.75) | 1.46 (0.67)
    Subscale 5 (finance): number analyzed (Participants) | 0 | 0 | 0 | 146 | 148 | 47 | 341
    Subscale 5 (finance) |  |  |  | 1.95 (0.89) | 1.83 (0.84) | 1.82 (0.83) | 1.88 (0.86)
PROMIS- Fatigue Number [Mean (Standard Deviation); unit: units on a scale] — Self report fatigue. Higher score= worse outcome. Population: Only caregivers reported outcome
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 146 | 148 | 47 | 341
    (all) |  |  |  | 2.29 (1.07) | 2.02 (1.00) | 2.38 (1.17) | 2.18 (1.06)

OUTCOME MEASURES:

1. Primary Outcome: Brief Fatigue Inventory (BFI)
Description: Aim 1: Average severity of fatigue over weeks 1-4 Individual Score Range: 0-10 Higher score means worse outcome
Time Frame: Week 1 -Week 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reflexology Patients | Meditative Practice Patients | Control Patients
Number analyzed (Participants) | 120 | 97 | 42
units on a scale | 4.17 (0.17) | 4.08 (0.18) | 4.32 (0.26)
Statistical Analysis 1: Comparison: Reflexology Patients vs Meditative Practice Patients; Aim 1: Comparing reflexology vs meditative practice for weeks 1-4; Test type: Superiority; p = .72, Mixed Models Analysis — Adjusted for baseline and balancing factors used in the randomization; Difference between least squared means = 0.09, 95% CI 2-sided [-.36 to .52] — Difference between reflexology and meditative practice for weeks 1-4
Statistical Analysis 2: Comparison: Reflexology Patients vs Control Patients; Aim 1: Comparing reflexology vs control for weeks 1-4; Test type: Superiority; p = .58, Mixed Models Analysis; Difference between least squared means = -0.15, 95% CI 2-sided [-.72 to .41] — Difference between reflexology and control for weeks 1-4
Statistical Analysis 3: Comparison: Meditative Practice Patients vs Control Patients; Aim 1: Comparing meditative practices vs control for weeks 1-4; Test type: Superiority; p = .42, Mixed Models Analysis; Difference between least squared means = -0.24, 95% CI 2-sided [-.81 to .34] — Difference between meditative practice and control for weeks 1-4

2. Primary Outcome: The MD Anderson Symptom Inventory (MDASI)- Distress
Description: Aim 1: Average severity of distress for weeks 1-4 Individual Score Range: 0-10 Higher score means worse outcome
Time Frame: Weeks 1-4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reflexology | Meditative Practice | Control
Number analyzed (Participants) | 120 | 97 | 42
units on a scale | 2.20 (0.17) | 2.21 (0.17) | 2.40 (0.25)
Statistical Analysis 1: Comparison: Reflexology vs Meditative Practice; Aim 1: Comparing reflexology vs meditative practice for weeks 1-4; Test type: Superiority; p = 0.96, Mixed Models Analysis; Difference between least squared means = -0.01, 95% CI 2-sided [-0.44 to 0.42] — Difference between reflexology and meditative practice for weeks 1-4
Statistical Analysis 2: Comparison: Reflexology vs Control; Aim 1: Comparing reflexology vs control for weeks 1-4; Test type: Superiority; p = 0.48, Mixed Models Analysis; Difference between least squared means = -0.2, 95% CI 2-sided [-0.75 to 0.35] — Difference between reflexology and control for weeks 1-4
Statistical Analysis 3: Comparison: Meditative Practice vs Control; Aim 1: Comparing meditative practice vs control for weeks 1-4; Test type: Superiority; p = 0.52, Mixed Models Analysis; Difference between least squared means = -0.19, 95% CI 2-sided [-0.75 to 0.38] — Difference between meditative practice and control for weeks 1-4

3. Primary Outcome: The MD Anderson Symptom Inventory (MDASI)- Summed Severity
Description: Aim 1: Average severity of symptoms from weeks 1-4 Summed range: 0-180 Higher score means worse outcome
Time Frame: Weeks 1-4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reflexology | Meditative Practice | Control
Number analyzed (Participants) | 120 | 97 | 42
units on a scale | 29.99 (1.27) | 29.32 (1.30) | 32.52 (1.87)
Statistical Analysis 1: Comparison: Reflexology vs Meditative Practice; Aim 1: Comparing reflexology vs meditative practice for weeks 1-4; Test type: Superiority; p = .68, Mixed Models Analysis; Difference between least squared means = 0.67, 95% CI 2-sided [-2.52 to 3.86] — Comparing reflexology to meditative practices for weeks 1-4
Statistical Analysis 2: Comparison: Reflexology vs Control; Aim 1: Comparing reflexology vs control for weeks 1-4; Test type: Superiority; p = .23, Mixed Models Analysis; Difference between least squared means = -2.53, 95% CI 2-sided [-6.64 to 1.58] — Comparing reflexology to control for weeks 1-4
Statistical Analysis 3: Comparison: Meditative Practice vs Control; Aim 1: Comparing meditative practice vs control for weeks 1-4; Test type: Superiority; p = 0.14, Mixed Models Analysis; Difference between least squared means = -3.2, 95% CI 2-sided [-7.41 to 1.01] — Comparing meditative practice to control for weeks 1-4

4. Primary Outcome: The MD Anderson Symptom Inventory (MDASI)- Sadness
Description: Aim 1: Average severity of sadness from weeks 1-4 Score range: 0-10 Higher score means worse outcome
Time Frame: Weeks 1-4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reflexology Patients | Meditative Practice Patients | Control Patients
Number analyzed (Participants) | 120 | 97 | 42
units on a scale | 1.79 (0.15) | 1.78 (0.16) | 2.03 (0.23)
Statistical Analysis 1: Comparison: Reflexology Patients vs Meditative Practice Patients; Aim 1: Comparing reflexology vs meditative practice for weeks 1-4; Test type: Superiority; p = 0.98, Mixed Models Analysis; Difference between least squared means = 0.01, 95% CI 2-sided [-0.38 to 0.39] — Difference between reflexology and meditative practice for weeks 1-4
Statistical Analysis 2: Comparison: Reflexology Patients vs Control Patients; Aim 1: Comparing reflexology vs control for weeks 1-4; Test type: Superiority; p = 0.34, Mixed Models Analysis; Difference between least squared means = -0.24, 95% CI 2-sided [-0.74 to 0.25] — Comparing reflexology to control for weeks 1-4
Statistical Analysis 3: Comparison: Meditative Practice Patients vs Control Patients; Aim 1: Comparing meditative practices vs control for weeks 1-4; Test type: Superiority; p = 0.34, Mixed Models Analysis; Difference between least squared means = -0.25, 95% CI 2-sided [-0.76 to 0.26] — Comparing meditative practices vs control for weeks 1-4

5. Secondary Outcome: Brief Fatigue Inventory (BFI)
Description: Aims 2 and 3: Average severity of fatigue for weeks 5-12 Score range: 0-10 Higher score means worse outcome
Time Frame: Weeks 5-12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Reflexology, Switching to Meditative Practices: Participants randomized into reflexology for weeks 1-4, then re-randomized to Meditative Practices for weeks 5-12
- Reflexology, Continuing With Reflexology: Participants randomized into reflexology for weeks 1-4 and continuing with reflexology for weeks 5-12
- Meditative Practice, Switching to Reflexology: Participants randomized to meditative practice for weeks 1-4, then re-randomized to reflexology for weeks 5-12
- Meditative Practice, Continuing With Meditative Practice: Participants randomized into meditative practice for weeks 1-4, then continued with meditative practice for weeks 5-12
Arm/Group | Reflexology, Switching to Meditative Practices | Reflexology, Continuing With Reflexology | Meditative Practice, Switching to Reflexology | Meditative Practice, Continuing With Meditative Practice
Number analyzed (Participants) | 32 | 36 | 27 | 30
units on a scale | 3.74 (0.38) | 3.99 (0.35) | 4.52 (0.52) | 4.03 (0.42)
Statistical Analysis 1: Comparison: Reflexology, Switching to Meditative Practices vs Reflexology, Continuing With Reflexology; Aim 2: After 4 weeks of reflexology, comparing continuing reflexology vs adding meditative practice; Test type: Superiority; p = 0.57, Mixed Models Analysis; Difference between least squared means = 0.25, 95% CI 2-sided [-.63 to 1.14] — After the initial 4 weeks of reflexology, comparing continued reflexology to added meditative practice
Statistical Analysis 2: Comparison: Meditative Practice, Switching to Reflexology vs Meditative Practice, Continuing With Meditative Practice; Aim 3: After 4 weeks of meditative practice, comparing continuing with meditative practice vs. adding reflexology for weeks 5-12; Test type: Superiority; p = 0.39, Mixed Models Analysis; Least Square (LS) Mean = 0.49, 95% CI 2-sided [-0.64 to 1.63] — After the initial 4 weeks of meditative practices, comparing continuing meditative practice to adding reflexology

6. Secondary Outcome: MD Anderson Symptom Inventory (MDASI)- Summed Severity
Description: Aims 2 and 3: Average severity of symptoms for weeks 5-12 Summed range: 0-180 Higher score means worse outcome
Time Frame: Weeks 5-12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reflexology, Switching to Meditative Practices | Reflexology, Continuing With Reflexology | Meditative Practice, Switching to Reflexology | Meditative Practice, Continuing With Meditative Practice
Number analyzed (Participants) | 27 | 32 | 21 | 29
units on a scale | 29.96 (3.97) | 28.02 (3.57) | 32.18 (3.76) | 30.33 (3.04)
Statistical Analysis 1: Comparison: Reflexology, Switching to Meditative Practices vs Reflexology, Continuing With Reflexology; Aim 2: After 4 weeks of reflexology, comparing continued reflexology vs added meditative practice for weeks 5-12; Test type: Superiority; p = 0.67, Mixed Models Analysis; Least Square (LS) Mean = 1.94, 95% CI 2-sided [-10.93 to 7.04] — After 4 weeks of reflexology, comparing continued reflexology vs adding meditative practice
Statistical Analysis 2: Comparison: Meditative Practice, Switching to Reflexology vs Meditative Practice, Continuing With Meditative Practice; Aim 3: After 4 weeks of meditative practices, comparing continued meditative practice vs adding reflexology for weeks 5-12; Test type: Superiority; p = 0.66, Mixed Models Analysis; Least Square (LS) Mean = -1.85, 95% CI 2-sided [-6.59 to 10.29] — After 4 weeks of meditative practice, comparing continued meditative practice vs adding reflexology for weeks 5-12

7. Secondary Outcome: MD Anderson Symptom Inventory (MDASI)- Distress
Description: Aims 2 and 3: Average severity of distress for weeks 5-12 Score range: 0-10 High score means worse outcome
Time Frame: Weeks 5-12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reflexology, Switching to Meditative Practices | Reflexology, Continuing With Reflexology | Meditative Practice, Switching to Reflexology | Meditative Practice, Continuing With Meditative Practice
Number analyzed (Participants) | 27 | 32 | 21 | 29
units on a scale | 2.28 (0.33) | 2.09 (0.30) | 2.11 (0.56) | 2.07 (0.48)
Statistical Analysis 1: Comparison: Reflexology, Switching to Meditative Practices vs Reflexology, Continuing With Reflexology; Aim 2: After 4 weeks of reflexology, comparing continued reflexology vs added meditative practice for weeks 5-12; Test type: Superiority; p = 0.62, Mixed Models Analysis; Difference between least squared means = -0.19, 95% CI 2-sided [-0.95 to 0.57] — After 4 weeks of reflexology, comparing continued reflexology vs added meditative practice for weeks 5-12
Statistical Analysis 2: Comparison: Meditative Practice, Switching to Reflexology vs Meditative Practice, Continuing With Meditative Practice; Aim 3: After 4 weeks of meditative practice, comparing continuing meditative practice vs adding reflexology for weeks 5-12; Test type: Superiority; p = 0.95, Mixed Models Analysis; Least Square (LS) Mean = -0.04, 95% CI 2-sided [-1.15 to 1.22] — After 4 weeks of meditative practice, comparing continued meditative practice vs adding reflexology for weeks 5-12

8. Secondary Outcome: MD Anderson Symptom Inventory (MDASI)- Sadness
Description: Aims 2 and 3: Average severity of sadness for weeks 5-12 Score range: 0-10 High score means worse outcome
Time Frame: Weeks 5-12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reflexology, Switching to Meditative Practices | Reflexology, Continuing With Reflexology | Meditative Practice, Switching to Reflexology | Meditative Practice, Continuing With Meditative Practice
Number analyzed (Participants) | 27 | 32 | 21 | 29
units on a scale | 2.17 (0.40) | 2.03 (0.36) | 2.01 (0.47) | 2.23 (0.38)
Statistical Analysis 1: Comparison: Reflexology, Switching to Meditative Practices vs Reflexology, Continuing With Reflexology; Aim 2: After 4 weeks of reflexology, comparing continued reflexology vs adding meditative practice for weeks 5-12; Test type: Superiority; p = 0.77, Mixed Models Analysis; Difference between least squared means = -0.14, 95% CI 2-sided [-1.04 to 0.77] — After 4 weeks of reflexology, comparing continued reflexology vs added meditative practice for weeks 5-12
Statistical Analysis 2: Comparison: Meditative Practice, Switching to Reflexology vs Meditative Practice, Continuing With Meditative Practice; Aim 3: After 4 weeks of meditative practice, comparing continued meditative practice vs added reflexology for weeks 5-12; Test type: Superiority; p = 0.67, Mixed Models Analysis; Least Square (LS) Mean = 0.22, 95% CI 2-sided [-1.23 to 0.80] — After 4 weeks of meditative practice, comparing continued meditative practice vs added reflexology for weeks 5-12

9. Secondary Outcome: Brief Fatigue Inventory (BFI)
Description: Aim 4: Average severity of fatigue for weeks 5-12 across initial 3 arms of study. The BFI instrument consists of nine items. The first three items ask respondents to rate the severity of fatigue "right now," at its "usual" level during the past 24 hours and at its "worst" level during the past 24 hours.
  Score range: 0-10 where 0 = no fatigue and 10 = as bad as you can imagine Higher score means worse outcome
Time Frame: Weeks 5-12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reflexology Patients | Meditative Practice Patients | Control Patients
Number analyzed (Participants) | 112 | 96 | 43
units on a scale | 3.62 (0.21) | 3.53 (0.21) | 3.87 (0.28)
Statistical Analysis 1: Comparison: Reflexology Patients vs Control Patients; Aim 4: Comparing reflexology vs control for weeks 5-12; Test type: Superiority; p = 0.42, Mixed Models Analysis; Least Square (LS) Mean = 0.09, 95% CI 2-sided [-0.88 to 0.37] — Comparing reflexology vs control for weeks 5-12
Statistical Analysis 2: Comparison: Meditative Practice Patients vs Control Patients; Aim 4: Comparing meditative practices vs control for weeks 5-12; Test type: Superiority; p = 0.29, Mixed Models Analysis; Least Square (LS) Mean = -0.34, 95% CI 2-sided [-0.98 to 0.29] — Comparing meditative practice vs control for weeks 5-12

10. Secondary Outcome: MD Anderson Symptom Inventory (MDASI)- Distress
Description: Aim 4: Average severity of distress for weeks 5-12 Score range: 0-10 Higher score means worse outcome
Time Frame: Weeks 5-12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reflexology Patients | Meditative Practice Patients | Control Patients
Number analyzed (Participants) | 112 | 96 | 43
units on a scale | 1.78 (0.19) | 2.00 (0.20) | 2.20 (0.26)
Statistical Analysis 1: Comparison: Reflexology Patients vs Control Patients; Aim 4: Comparing reflexology vs control for weeks 5-12; Test type: Superiority; p = 0.15, Mixed Models Analysis; Least Square (LS) Mean = -0.42, 95% CI 2-sided [-1.00 to 0.15] — Comparing reflexology vs control for weeks 5-12
Statistical Analysis 2: Comparison: Meditative Practice Patients vs Control Patients; Aim 4: Comparing meditative practice vs control for weeks 5-12; Test type: Superiority; p = 0.50, Mixed Models Analysis; Least Square (LS) Mean = -0.2, 95% CI 2-sided [-0.80 to 0.39] — Comparing meditative practice vs control for weeks 5-12

11. Secondary Outcome: MD Anderson Symptom Inventory (MDASI)- Sadness
Description: Aim 4: Average severity of sadness for weeks 5-12 Score range: 0-10 Higher score means worse outcome
Time Frame: Weeks 5-12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reflexology Patients | Meditative Practice Patients | Control Patients
Number analyzed (Participants) | 112 | 96 | 43
units on a scale | 1.75 (0.18) | 1.66 (0.19) | 2.02 (0.25)
Statistical Analysis 1: Comparison: Reflexology Patients vs Control Patients; Aim 4: Comparing reflexology vs control for weeks 5-12; Test type: Superiority; p = 0.33, Mixed Models Analysis; Least Square (LS) Mean = -0.27, 95% CI 2-sided [-0.83 to 0.28] — Comparing reflexology vs control for week 5-12
Statistical Analysis 2: Comparison: Meditative Practice Patients vs Control Patients; Aim 4: Comparing meditative practice vs control for weeks 5-12; Test type: Superiority; p = 0.22, Mixed Models Analysis; Least Square (LS) Mean = -0.36, 95% CI 2-sided [-0.93 to 0.21]

12. Secondary Outcome: MD Anderson Symptom Inventory (MDASI)- Summed Severity
Description: Aim 4: Comparing average severity of symptoms for weeks 5-12 Summed score range: 0-180 Higher score means worse outcome
Time Frame: Weeks 5-12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Meditative Practive Patients: Patients randomized into the meditative practice arm, given meditative practice from a friend/ family member.
  Meditative Practices include elements of meditation, gentle yoga and breathing exercises. These practices focus purposeful attention to the present moment and have been shown to enhance one's ability to adapt to serious health concerns
Arm/Group | Reflexology Patients | Meditative Practive Patients | Control Patients
Number analyzed (Participants) | 112 | 96 | 43
units on a scale | 26.69 (1.66) | 25.77 (1.70) | 30.25 (2.28)
Statistical Analysis 1: Comparison: Reflexology Patients vs Control Patients; Aim 4: Comparing reflexology vs control for weeks 5-12; Test type: Superiority; p = 0.17, Mixed Models Analysis; Least Square (LS) Mean = 0.92, 95% CI 2-sided [-8.62 to 1.52] — Comparing reflexology vs control for weeks 5-12
Statistical Analysis 2: Comparison: Meditative Practive Patients vs Control Patients; Aim 4: Comparing meditative practice vs control for weeks 5-12; Test type: Superiority; p = 0.09, Mixed Models Analysis; Least Square (LS) Mean = -4.48, 95% CI 2-sided [-9.66 to 0.70] — Comparing meditative practice vs control for weeks 5-12

ADVERSE EVENTS:
Time Frame: Data was collected over 12 weeks
Arm/Group | Reflexology | Meditative Practice | Control
All-Cause Mortality (participants affected / at risk) | 4/150 | 5/150 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150 | 0/47
Other Adverse Events (participants affected / at risk) | 0/150 | 0/150 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT02759146/Prot_SAP_000.pdf